CLINICAL TRIAL: NCT02668016
Title: Self-Assessment Method for Statin Side-effects Or Nocebo
Acronym: SAMSON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 15SM2947; 2015-004109-18 (EudraCT Number)
Record Dates: First submitted 2016-01-19; First posted 2016-01-29 (Estimated); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Adverse Effects; Cardiovascular Diseases; Hyperlipidemias
Keywords: cardiovascular diseases; hyperlipidemias
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atorvastatin 20mg Daily (Experimental): Atorvastatin 20mg daily for 1 month
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Placebo daily for 1 month
  Interventions: Other: Placebo
- No Treatment (No Intervention): No Atorvastatin or placebo for 1 month

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 20mg tablets taken orally once daily for one month.
  Other Names: HMG CoA reductase inhibitors; Statins
  Arms: Atorvastatin 20mg Daily
Other: Placebo — Placebo tablets taken orally once daily for one month
  Arms: Placebo

SUMMARY:
Front-line clinicians cannot currently test for an individual participant whether symptoms experienced are the pharmacological result of a statin or due to other phenomena. In this trial, participants who have previously ceased statins due to side effects will be offered the opportunity to undergo twelve randomly ordered 1-month periods. There will be four periods of no medication, four periods of placebo and four periods of statin. The placebo and the statin pills will be identical in appearance. Participants will record on a daily basis side-effects experienced. At the end of the study, the one-month sessions are sorted into the order shown above. The participant can then observe directly how much of the increase in symptoms seen with statin is also seen with placebo.

1. Hypothesis 1: that >30% of participants enrolling for the study will complete it.
2. Hypothesis 2: Overall >50% of symptom burden is nocebo rather than pharmacological
3. The investigators will define the Nocebo proportion of side effects.
4. Hypothesis 3: that the majority of participants, at 6 months after completion, will either be taking statins or have declined statins for reasons other than perceived side effects.

DETAILED DESCRIPTION:
Participants: 50 participants will be recruited to the trial.

Method: At baseline each participant will have a detailed interview with the study doctor to assess past medical history and previous symptoms attributed to statins and assess if they are eligible to be enrolled. Eligible participants will be enrolled and allocated a random predefined order to take the study interventions in. These random codes will be generated by the trials unit statistician and supplied to the production pharmacy. The participant will be dispensed High Density Polyethylene (HDPE) containers which are in this pre-specified order. Each participant will receive 12 sets of HDPE containers pre-labelled. 4 sets of HDPE containers will contain no medication, 4 will contain 1-month supply of matched placebo and 4 will contain 1-month supply of atorvastatin 20mg. At the start of the next calendar month after the screening visit the participants will commence the trial intervention. The research nurse will call the participant to remind them to start on the 1st day of the next month after screening. Each day participants will rate their daily symptom on a phone application and will also complete 3 additional questionnaires on a monthly basis. The study nurse will call the participant at the end of each month to assess their progress in the trial. Each participant will return their boxes at dispensing visits (if applicable) and at the study end in order for a pill count to be undertaken to assess medication adherence. The placebo and atorvastatin pills will be visually identical.

The study enrols participants not intending to re-start clinical use of statins. Participants' other medications will continue to be managed as normal by their own physicians, with no restriction on starting, stopping or changing doses. For safety reasons the participant's own physician will be asked to consult the investigators prior to consideration of starting, or amending the dose of, any other lipid lowering medication.

For the trial, each participant will receive a smartphone, or if preferred, can have the application downloaded to their existing phone to allow real-time daily documentation of symptoms experienced on a visual analogue scale of 0-100. Participants will receive training on the simple touch-screen interface and a leaflet with further information will also be provided. Participants will rate symptoms every day, with the daily scores aggregated into a monthly score. This is preferable over scoring only once a month, because participants may struggle to remember and aggregate their symptom burden especially if it varies between days.

Each month participants will fill out two validated questionnaires on the impact of their side-effects on their quality of life. These are EuroQol (EQ-5D-3L), a well-validated measure of health related quality of life, and the Treatment Satisfaction Questionnaire for Medicine (TSQM) questionnaire, a validated treatment satisfaction questionnaire. EQ-5D-3L assesses five domains of health and overall self-rated health using a visual analogue scale. EQ-5D-3L is conventional for assessing efficacy of medication on quality of life but may not be sufficient for assessing side effects, therefore the TSQM questionnaire will also be used. Use of both a health related quality of life questionnaire and a treatment satisfaction questionnaire will allow assessment of participants' multiple health states, overall self-rated health status and treatment satisfaction, and provide a test of both convergent validity and measurement invariance for the monthly aggregate symptom burden score.

The investigators will also ask participants to fill in a short questionnaire detailing any potentially their own physicians, with no restriction on starting, stopping or changing doses For safety reasons the participant's own physician will be asked to consult the investigators prior to consideration of starting, or amending the dose of, any other lipid lowering medication.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Previously taken one or more statins
* Withdrawn from statins because of perceived side effects
* Developed side effects within 2 weeks of initiation
* Clinical indication for statins for primary or secondary prevention of cardiovascular disease or dyslipidaemia, on either no medication or non-statin lipid lowering therapy (e.g, ezetimibe)

Exclusion Criteria:

* History of neuropathy
* Regularly taking prescribed analgesia
* History of a chronic pain condition
* History of severe mental illness (as their experience of symptoms may already be altered)
* Current use of fibrates (because of the risk of interaction with statins; will not exclude participants taking ezetimibe).
* Severe previous reaction or reaction considered immunological, such as anaphylaxis, facial swelling, severe rash, muscle ache with rise in serum creatine kinase, inflammatory myopathy, rhabdomyolysis or liver function abnormalities (aspartate transaminase (AST) or alanine transaminase (ALT) greater than 3 times upper limit or normal).
* Side-effects taking longer than 2 weeks to develop (because in such participants much longer blocks of treatment would be required; if the present study is positive such studies will be planned for the future).
* History of statin intolerance with drug interaction to antiretroviral drugs.
* Currently taking antiretrovirals with known interaction to statins
* Currently taking any drug other than antiretrovirals with known interaction to statins
* Side effects taking longer than 2 weeks to present.
* In clinical judgement of study doctor, participant should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrel P Francis, MB MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howard JP, Wood FA, Finegold JA, Nowbar AN, Thompson DM, Arnold AD, Rajkumar CA, Connolly S, Cegla J, Stride C, Sever P, Norton C, Thom SAM, Shun-Shin MJ, Francis DP. Side Effect Patterns in a Crossover Trial of Statin, Placebo, and No Treatment. J Am Coll Cardiol. 2021 Sep 21;78(12):1210-1222. doi: 10.1016/j.jacc.2021.07.022. PMID 34531021

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All participants received:
  Atorvastatin 20mg daily taken orally for one month or placebo daily for one month or no tablets for one month.
  Each participant was randomised to 4 x 1-month periods of Atorvastatin 20mg daily taken orally for one month and 4 x 1-month periods of placebo daily for one month and 4 x 1 no tablets daily for one month.
  The 12 treatment periods could be in any order.
Period: Month 1
Arm/Group | All Study Participants
Started | 60
Received Atorvastatin 20mg | 20
Received Placebo | 20
Received No Tablet | 20
Withdrew | 0
Completed | 55
Not Completed | 5
Period: Month 2
Arm/Group | All Study Participants
Started | 60
Received Atorvastatin 20mg | 20
Received Placebo | 20
Received No Tablet | 20
Withdrew | 2
Completed | 54
Not Completed | 6
Not completed — Withdrew due to other health condition preventing continuation with the protocol | 1
Not completed — Withdrew due to repeated failure to provide treatment scores | 1
Not completed — Not applicable - stopped trial medication for rest of month but continued in the trial | 4
Period: Month 3
Arm/Group | All Study Participants
Started | 58
Received Atorvastatin 20mg | 18
Received Placebo | 20
Received No Tablet | 20
Withdrew | 0
Completed | 47
Not Completed | 11
Period: Month 4
Arm/Group | All Study Participants
Started | 58
Received Atorvastatin 20mg | 19
Received Placebo | 19
Received No Tablet | 20
Withdrew | 2
Completed | 53
Not Completed | 5
Not completed — Withdrawal due to severe symptoms | 1
Not completed — Withdrawal due to non-compliance with trial protocol | 1
Not completed — Not applicable - stopped trial medication for rest of month but continued in the trial | 3
Period: Month 5
Arm/Group | All Study Participants
Started | 56
Received Atorvastatin 20mg | 18
Received Placebo | 19
Received No Tablet | 19
Withdrew | 0
Completed | 53
Not Completed | 3
Period: Month 6
Arm/Group | All Study Participants
Started | 56
Received Atorvastatin 20mg | 19
Received Placebo | 17
Received No Tablet | 20
Withdrew | 4
Completed | 50
Not Completed | 6
Not completed — Withdrawal as decided side effects non longer statin mediated | 1
Not completed — Withdrawal due to severe symptoms | 2
Not completed — Withdrawal due to other health issues preventing continuation with the protocol | 1
Not completed — Not applicable - stopped trial medication for rest of month but continued in the trial | 2
Period: Month 7
Arm/Group | All Study Participants
Started | 52
Received Atorvastatin 20mg | 18
Received Placebo | 18
Received No Tablet | 16
Withdrew | 0
Completed | 43
Not Completed | 9
Period: Month 8
Arm/Group | All Study Participants
Started | 52
Received Atorvastatin 20mg | 18
Received Placebo | 19
Received No Tablet | 15
Withdrew | 1
Completed | 45
Not Completed | 7
Not completed — Withdrawal due to severe symptoms | 1
Not completed — Not applicable - stopped trial medication for rest of month but continued in the trial | 6
Period: Month 9
Arm/Group | All Study Participants
Started | 51
Received Atorvastatin 20mg | 15
Received Placebo | 19
Received No Tablet | 17
Withdrew | 0
Completed | 40
Not Completed | 11
Period: Month 10
Arm/Group | All Study Participants
Started | 51
Received Atorvastatin 20mg | 15
Received Placebo | 18
Received No Tablet | 18
Withdrew | 2
Completed | 43
Not Completed | 8
Not completed — Withdrawal due to intercurrent social stresses | 1
Not completed — Withdrawal due to severe symptoms | 1
Not completed — Not applicable - stopped trial medication for rest of month but continued in the trial | 6
Period: Month 11
Arm/Group | All Study Participants
Started | 49
Received Atorvastatin 20mg | 17
Received Placebo | 15
Received No Tablet | 17
Withdrew | 0
Completed | 42
Not Completed | 7
Period: Month 12
Arm/Group | All Study Participants
Started | 49
Received Atorvastatin 20mg | 16
Received Placebo | 17
Received No Tablet | 16
Withdrew | 0
Completed | 43
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Crossover design
Groups:
- Atorvastatin 20mg Daily: Atorvastatin 20mg daily for 1 month or Placebo daily or No Treatment
Arm/Group | Atorvastatin 20mg Daily
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Symptom Scores Across Statin, Placebo and no Treatment Periods
Description: The full scale name would be "daily symptom score" measuring patient-reported symptoms on a scale from 0 (no symptoms) to 100 (worst imaginable symptoms). The unit of measurement would be "scores on a scale".
  The mean symptom scores for the four months on each arm will be calculated: placebo, Atorvastatin 20mg and no treatment. Mean symptom scores across statin, placebo and no treatment periods is calculated. There are no subscales/subranges.
Time Frame: 12 months
Population: Crossover trial - The primary end point was symptom intensity as assessed with the use of the nocebo ratio (i.e., the ratio of symptom intensity induced by taking placebo to the symptom intensity induced by taking a statin). This ratio was calculated as the symptom intensity with placebo minus the symptom intensity with neither statin nor placebo, divided by the symptom intensity with a statin minus the symptom intensity with neither statin nor placebo.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atorvastatin 20mg Daily | Placebo | No Treatment
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 16.3 [13.0 to 19.6] | 15.4 [12.1 to 18.7] | 8.0 [4.7 to 11.3]

2. Secondary Outcome: Number of Participants Currently Being Prescribed Statins
Description: Following the end of the trial, is the trial participant taking statins or not.
Time Frame: At 6-months after the end of trial up to 7-months
Population: Cross-over design
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 20mg Daily | Placebo | No Treatment
Number analyzed (Participants) | 60 | 0 | 0
Participants | 30 | 0 | 0

3. Secondary Outcome: Attribution of Adverse Symptoms
Description: Following the end of the trial, whether individual trial participants currently believe that most of the side-effects previously attributed to the statin, were indeed a pharmacological effect of the statin.
Time Frame: 6-months after end of trial
Measure: Number; unit: participants
Groups:
- Attribution of Side Effects 6-months After End of Trial: Following the end of the trial, whether individual trial participants currently believe that most of the side-effects previously attributed to the statin, were indeed a pharmacological effect of the statin.
Arm/Group | Attribution of Side Effects 6-months After End of Trial
Number analyzed (Participants) | 60
participants
  Yes | 22
  No | 17
  Unknown | 8
  Other | 3
  Undecided | 9
  Lost to follow-up | 1

ADVERSE EVENTS:
Time Frame: 12-months of the trial and for six-months post-trial until the participant had completed their end of study plus six-month visit.
Description: Definition of adverse events does not differ to clinicaltrials.gov.
Groups:
- In-Follow-up: Completed or withdrawn from trial intervention but in follow-up until end of trial +6-month follow-up visit.
Arm/Group | Atorvastatin 20mg Daily | Placebo | No Treatment | In-Follow-up
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 5/60 | 3/60 | 1/60 | 10/60
Other Adverse Events (participants affected / at risk) | 36/60 | 42/60 | 23/60 | 6/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin 20mg Daily (N=60) | Placebo (N=60) | No Treatment (N=60) | In-Follow-up (N=60)
Polycythemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Obstructive Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Hemoperitoneum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast Cancer (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Cardiopulmonary bypass (Surgical and medical procedures) | 0 | 0 | 0 | 1
Shoulder Arthroplasty (Surgical and medical procedures) | 1 | 1 | 1 | 1
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Transient Ischaemic Attack (Vascular disorders) | 0 | 0 | 0 | 1
Myocardial Infarction (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin 20mg Daily (N=60) | Placebo (N=60) | No Treatment (N=60) | In-Follow-up (N=60)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (39) | 23 (33) | 3 (3) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 15 (19) | 9 (12) | 1 (1)
Fatigue (General disorders) | 10 (13) | 12 (15) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (14) | 6 (6) | 2 (2) | 3 (3)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (11) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 7 (7) | 5 (6) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (9) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 4 (4) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 3 (3) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
To be eligible for the trail, patients' previous perceived side effects whilst taking statins must have arisen within 2 weeks of commencing the drug. This is to ensure the 1 month long blocks are long enough that symptoms would be expected to arise.

Patients whose symptoms take longer than 2 weeks to arise were not eligible for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT02668016/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT02668016/SAP_001.pdf